CLINICAL TRIAL: NCT01860729
Title: A 24-Week, Worldwide, Multicenter, Double-Blind, Randomized, Parallel, Placebo- Controlled Study to Assess the Efficacy and Tolerability of Anacetrapib When Added to Ongoing Statin Therapy With or Without Other Lipid Modifying Medication(s) in Patients With Hypercholesterolemia or Low HDL-C
Brief Title: A Study of the Safety and Efficacy of Anacetrapib (MK-0859) Among Participants With Hypercholesterolemia When Added to Ongoing Statin Therapy (MK-0859-022)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0859-022
Record Dates: First submitted 2013-05-20; First posted 2013-05-23 (Estimated); Last update posted 2020-05-29 (Actual); Status verified 2020-05

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — anacetrapib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Anacetrapib (Experimental): 100 mg tablet, oral, once daily for 24 weeks
  Interventions: Drug: Anacetrapib
- Placebo (Placebo Comparator): Matching tablet to Anacetrapib 100 mg, oral, once daily for 24 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Anacetrapib
  Other Names: MK-0859
  Arms: Anacetrapib
Drug: Placebo
  Arms: Placebo

SUMMARY:
This study will evaluate the effects of anacetrapib on low-density lipoprotein-cholesterol (LDL-C) and high-density lipoprotein cholesterol (HDL-C) in participants with hypercholesterolemia when added to an existing statin therapy.

ELIGIBILITY:
Inclusion Criteria:

* If female, cannot be of reproductive potential
* Has been treated with an appropriate dose of statin for at least 6 weeks
* Coronary heart disease (CHD) or other atherosclerotic vascular disease with multiple risk factors (including diabetes, metabolic syndrome) and/or high LDL-C/low HDL-C, or needing to meet a specific LDL-C/HDL-C goal

Exclusion Criteria:

* Previously participated in a study with a cholesteryl ester transfer protein (CETP) inhibitor
* Homozygous familial hypercholesterolemia
* Severe chronic heart failure
* Uncontrolled cardiac arrhythmias, myocardial infarction (MI), percutaneous coronary intervention (PCI), coronary artery by-pass graft (CABG), unstable angina, or stroke within 3 months
* Uncontrolled hypertension
* Uncontrolled endocrine or metabolic disease known to influence serum lipids or lipoproteins
* Active or chronic hepatobiliary, hepatic, or gall bladder disease
* History of mental instability, drug/alcohol abuse within the past five years or major psychiatric illness inadequately controlled and unstable
* History of ileal bypass, gastric bypass, or other significant condition associated with malabsorption
* Human immunodeficiency virus (HIV) positive
* History of malignancy ≤5 years
* Donated blood products or has had phlebotomy of >300 mL within 8 weeks or intends to donate 250 mL of blood products or receive blood products within the projected duration of the study
* Currently taking medications that are potent inhibitors or inducers of cytochrome P450 3A4 (CYP3A) (including but not limited to cyclosporine, systemic itraconazole or ketoconazole, erythromycin, clarithromycin, or telithromycin, nefazodone, protease inhibitors, carbamazepine, phenobarbital, phenytoin, rifabutin, rifampin, St John's wort) or has discontinued treatment <3 weeks prior
* Consumes more than 2 alcoholic drinks per day
* Currently participating or has participated in a study with an investigational compound or device within 3 months
* Receiving treatment with systemic corticosteroids or taking systemic anabolic agents

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 589 (Actual)
Dates: Start 2013-05-13 (Actual); Primary Completion 2015-05-29 (Actual); Study Completion 2015-08-20 (Actual)

PRIMARY OUTCOMES:
Percent Change from Baseline in LDL-C (beta-quantification [BQ] method) | Baseline and Week 24
Percent Change from Baseline in HDL-C | Baseline and Week 24
Number of Participants with Alanine Transaminase (ALT) or Aspartate Aminotransferase (AST) Consecutive Elevations ≥3x Upper Limit of Normal (ULN) | 24 weeks
Number of Participants with Creatine Phosphokinase Elevations ≥10xULN with or without Muscle Symptoms | 24 weeks
Number of Participants with Sodium, Chloride, or Bicarbonate Elevations >ULN or Potassium Levels <Lower Limit of Normal (LLN) | 24 weeks
Number of Participants with Pre-specified Adjudicated Cardiovascular Serious Adverse Events or Death from Any Cause | 24 weeks
Number of Participants with Significant Increase in Blood Pressure | 24 weeks

SECONDARY OUTCOMES:
Percent Change from Baseline in non-HDL-C | Baseline and Week 24
Percent Change from Baseline in Apolipoprotein B (Apo-B) | Baseline and Week 24
Percent Change from Baseline in Apolipoprotein A-I (Apo-A-I) | Baseline and Week 24
Percent Change from Baseline in Lipoprotein(a) (lp[a]) | Baseline and Week 24
Percent Change from Baseline in HDL-C Among Participants with Low HDL-C at LDL-C Goal | Baseline and Week 24

REFERENCES:
- [Result] Ballantyne CM, Shah S, Sapre A, Ashraf TB, Tobias SC, Sahin T, Ye P, Dong Y, Sheu WH, Kang DH, Ferreira Rossi PR, Moiseeva Y, Briones IR, Johnson-Levonas AO, Mitchel YB. A Multiregional, Randomized Evaluation of the Lipid-Modifying Efficacy and Tolerability of Anacetrapib Added to Ongoing Statin Therapy in Patients With Hypercholesterolemia or Low High-Density Lipoprotein Cholesterol. Am J Cardiol. 2017 Aug 15;120(4):569-576. doi: 10.1016/j.amjcard.2017.03.255. Epub 2017 Apr 12. PMID 28624096